CLINICAL TRIAL: NCT02871401
Title: A Phase One-B (1B) Pilot Trial of Herpesvirus Treatment in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Pilot Trial of Herpesvirus Treatment in Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Kropski, Assistant Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160693
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Herpesvirus; Valganciclovir
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Herpes Simplex | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valganciclovir (Experimental): Valganciclovir 450 mg, 2 pills by mouth one time per day x 12 weeks
  Interventions: Drug: Valganciclovir
- Placebo (Placebo Comparator): Placebo, 2 pills by mouth one time per day x 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valganciclovir — Subjects with IPF currently tolerating pirfenidone treatment who have evidence of prior EBV or CMV infection will be randomized to valganciclovir or placebo for 12 weeks.
  Other Names: Valcyte
  Arms: Valganciclovir
Drug: Placebo — Subjects with IPF currently tolerating pirfenidone treatment who have evidence of prior EBV or CMV infection will be randomized to valganciclovir or placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
The investigators will conduct a single-center, prospective, randomized, placebo-controlled, double-blind pilot study of anti-herpesvirus therapy in patients with idiopathic pulmonary fibrosis (IPF). Patients with mild, moderate or severe IPF with serologic evidence of current or past Epstein-Barr Virus (EBV) or cytomegalovirus (CMV) infection. Randomization will be to pirfenidone plus placebo or pirfenidone plus valganciclovir. Thirty subjects will be enrolled and randomized to treatment with pirfenidone plus valganciclovir (20 subjects) or pirfenidone plus placebo (10 subjects) for 12 weeks. The primary outcome will be safety and tolerability will be determined by type, frequency and duration of adverse events (AEs) and serious adverse events (SAEs) after 12 weeks of study drug treatment. All study subjects will be offered bronchoscopy with bronchoalveolar lavage (BAL) at study initiation and upon completion of treatment (12 weeks). Subjects will then be followed up at routine clinic visits at 6, 9 and 12 months for data collection.

ELIGIBILITY:
Inclusion Criteria:

1. age >21 and <80 years
2. ability to provided informed consent
3. diagnosis of probable or definite IPF according to American Thoracic Society (ATS) criteria
4. tolerance of full-dose (2403 mg/day) pirfenidone
5. Positive serology for EBV or CMV

Exclusion Criteria:

1. FVC < 40% predicted
2. Diffusing capacity for carbon monoxide (DLCO) < 35% predicted (Crapo)
3. Forced expiratory volume (FEV)1/FVC <0.7
4. Significant centrilobular emphysema (>40% by HRCT)
5. Active tobacco use (cigarette or cigar smoking)
6. Resting oxygen saturation (SpO2) on room air <89%
7. Listed for lung transplantation defined as being assigned a lung allocation score
8. environmental exposure (occupational, environmental, drug, etc.) felt by the principal investigator (PI) to be the etiology of the interstitial disease
9. diagnosis of collagen-vascular conditions (according to the published American College of Rheumatology criteria)
10. history of unstable or deteriorating cardiac disease
11. acute coronary syndrome, coronary artery bypass, or angioplasty within 3 months of screening
12. uncontrolled arrhythmia
13. uncontrolled hypertension
14. known HIV or hepatitis C
15. known cirrhosis or chronic active hepatitis
16. active substance or alcohol abuse
17. pregnancy or lactation
18. Women of childbearing potential who are not using a medically approved means of contraception. Subjects will be considered of childbearing potential if they are not surgically sterile or have not been postmenopausal for at least 2 years [any subject who is postmenopausal for < 2 years will be required to have a follicle-stimulating hormone (FSH) level to assess her potential to become pregnant
19. clinically relevant lab abnormalities (obtained within 30 days before enrollment), including:

    1. creatinine > 2 x upper limit of normal (ULN)
    2. hematology outside of specified limits: white blood cells (WBCs) < 3,500/mm3; hematocrit < 25% or > 59%; platelets < 100,000/mm3;
    3. total bilirubin > 2 x ULN
    4. Aspartate (AST) or alanine aminotransferases (ALT)/ serum glutamic-oxaloacetic; transaminase (SGOT), or serum glutamic pyruvic transaminase (SGPT) > 2.0 x ULN
    5. alkaline phosphatase > 3 x ULN
    6. albumin < 3.0 mg/dL at screening
20. known hypersensitivity to study medication
21. any condition that, in the judgment of the PI, might cause participation in this study to be detrimental to the subject or that the PI deems makes the subject a poor candidate
22. any therapy with immunosuppressants such as prednisone, azathioprine, or mycophenolate currently or anticipated to be needed during the study period (subjects on these drugs prior to the study will require a 30-day washout period before randomization)
23. participation in another IPF clinical treatment trial during the study period (if completing another IPF clinical treatment trial, then a 30-day washout period is required before randomization)
24. requirement for chronic suppressive therapy with valacyclovir for recurrent herpes virus infection
25. History of myelodysplasia, aplastic anemia, refractory anemia, or multiple myeloma.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Kropski, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Blackwell TS, Hewlett JC, Mason WR, Martin S, Del Greco J, Ding G, Wu P, Lancaster LH, Loyd JE, Dudenhofer RB, Salisbury ML, Kropski JA. A Phase I Randomized, Controlled, Clinical Trial of Valganciclovir in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2021 Aug;18(8):1291-1297. doi: 10.1513/AnnalsATS.202102-108OC. PMID 33740394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valganciclovir | Placebo
Started | 20 | 11
Completed | 19 | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valganciclovir | Placebo | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (6.8) | 68.8 (8.0) | 68.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 16 | 9 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 11 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 11 | 31
Forced vital capacity (FVC) % predicted for age [Mean (Standard Deviation); unit: %] | 69.4 (19.0) | 69.4 (7.7) | 69.4 (15.8)
Forced expiratory volume in 1 second (FEV1) % predicted for age [Mean (Standard Deviation); unit: %] | 76.9 (20.5) | 79.7 (10.8) | 77.9 (17.5)
Total Lung Capacity (TLC) % predicted for age [Mean (Standard Deviation); unit: %] | 62.2 (17.7) | 62.1 (7.2) | 62.2 (14.4)
Diffusion capacity for carbon monoxide (DLCO) % predicted for age [Mean (Standard Deviation); unit: %] | 47.3 (10.2) | 41.0 (8.9) | 45.0 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Discontinue Study Drug Due to Adverse Events
Description: Proportion of study subjects who discontinue study drug due to adverse events
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 20 | 11
Participants | 1 | 0

2. Secondary Outcome: Adverse Events - Number
Description: Number of subjects with each reported adverse event
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 20 | 11
participants
  At least 1 AE | 14 | 4
  Cough | 3 | 1
  Leukocytosis | 1 | 3
  Diarrhea | 2 | 0
  Elevated liver enzymes | 2 | 0
  Pneumonia | 2 | 0
  Worsened dyspnea | 0 | 2
  Acute pain of shoulder | 1 | 0
  Acute respiratory failure | 1 | 0
  Acute sinusitis | 1 | 0
  Bilateral arm swelling | 1 | 0
  Bilateral lower leg edema | 1 | 0
  Carbuncle on face | 1 | 0
  Depression | 0 | 1
  Dyspepsia | 0 | 1
  Hoarseness | 0 | 1
  Hypertension | 0 | 1
  Hypoxia during flight | 0 | 1
  Jaw pain | 0 | 1
  Lymphopenia | 1 | 0
  Nausea | 0 | 1
  Nephrolithiasis | 1 | 0
  Pain in back | 0 | 1
  Paroxysmal atrial fibrillation | 1 | 0
  Prostate cancer recurrence | 0 | 1
  Rash | 1 | 0
  Respiratory tract infection | 1 | 0
  Sore throat | 1 | 1
  Thrombocytopenia | 1 | 0
  Tooth pain | 1 | 0
  Upper respiratory tract infection | 1 | 0
  Vertigo | 1 | 0
  Weakness | 1 | 0
  Weight loss | 1 | 0
  Worsening anemia | 0 | 1
  Worsening hypertension | 1 | 0

3. Secondary Outcome: Serious Adverse Events
Description: Number of subjects with each serious adverse event
Time Frame: 12 weeks
Population: Serious adverse events
Measure: Number; unit: events
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 20 | 11
events | 2 | 1

4. Secondary Outcome: Total # Adverse Events
Description: Total number of adverse events
Time Frame: Randomization to 16 weeks
Measure: Number; unit: events
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 20 | 11
events | 33 | 13

5. Other Pre Specified Outcome: Change in Forced Vital Capacity (FVC)
Description: Change in FVC percent predicted compared to baseline
Time Frame: Baseline vs. 12 weeks, 1 year
Population: PFT data not available at 1 year (obtained per standard of-care at clinical visit) for 5 subjects.
  Reasons for missing data: Decreased (n=1), moved out of region and lost to follow-up (n=1), PFT's not obtained at visit (n=3).
Measure: Median (Inter-Quartile Range); unit: percentage predicted
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 20 | 11
percentage predicted
  Baseline to 12 weeks | 0 [-1 to 2] | -2 [-4 to 2]
  Baseline to 12 months: number analyzed (Participants) | 19 | 7
  Baseline to 12 months | -1 [-4 to 1] | -5 [-10 to 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through active treatment (week 12) and 4 weeks of additional follow-up.
Description: AE's were assessed by study personnel at each study visit.
Arm/Group | Valganciclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/11
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/11
Other Adverse Events (participants affected / at risk) | 14/20 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valganciclovir (N=20) | Placebo (N=11)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Diffuse skin rash
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonia
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valganciclovir (N=20) | Placebo (N=11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bilateral upper extremity edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BIlateral lower extremity edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hoarseness (General disorders) | 1 (1) | 0 (0)
Hypoxia during flight (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Jaw pain (General disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain in back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sore throat (General disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tooth pain (General disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Worsening hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT02871401/Prot_SAP_000.pdf